CLINICAL TRIAL: NCT00161291
Title: A Phase II Open Label Trial of Pre-Operative (Neoadjuvant) Letrozole in Combination With Bevacizumab in Post-Menopausal Women With Newly Diagnosed Operable Breast Cancer
Brief Title: Open Label Trial for Post-Menopausal Women With Newly Diagnosed Operable Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Andres Forero, M.D., UAB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F041222006; UAB 0467 (Other: Institutional protocol study number)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer
Keywords: Carcinoma of the breast; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Letrozole in combination with Bevacizumab — Patients will be administered Letrozole at 2.5 mg PO a day and Avastin at 15 mg/kg IV every 3 weeks for 24 weeks. Patients will then undergo surgical treatment and receive adjuvant therapy according to the treating physician.
  Other Names: Letrozole (Femara); Bevacizumab (Avastin)

SUMMARY:
The purpose of this study is to determine pathological response to a maximum of 18 weeks of neoadjuvant therapy using a combination of letrozole and Bevacizumab in post-menopausal women with pathologically confirmed invasive ductal cancer or invasive lobular cancer of the breast whose tumors are hormone positive.

DETAILED DESCRIPTION:
This is an open label, single arm, and Phase II study of the combination of Letrozole and Bevacizumab in patients with newly diagnosed breast cancer. Patients meeting the eligibility criteria and who have signed the consent form will start Letrozole 2.5 mg by mouth a day and Bevacizumab 15 mg per Kg IV every 3 weeks for 18 weeks (24 weeks if still responding at week 18 if approved by the PI). After neoadjuvant therapy, participants will undergo surgical treatment and will receive adjuvant therapy according to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive ductal carcinoma or invasive lobular carcinoma of the breast, T2-T4 / T4a-c / N0-2 / M0, with positive estrogen and/or progesterone receptors. Patients with inflammatory breast cancer will not be included (Stage IIIb). Patients previously treated patients with no measurable disease or patients with metastatic disease will be excluded.
* Written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice (see Appendix B - consent form).
* Females 60 years of age (postmenopausal).
* Be ambulatory (outpatient) and have an ECOG PS <2 (Appendix F).
* Patients must have measurable disease by mammogram and/or breast ultrasound. The target lesion must not have been previously irradiated.
* No prior chemotherapy.
* Patients must have adequate organ and marrow function as defined as follows: absolute neutrophil count > 1,500/mm3, hemoglobin > 8.0 g/dl, platelets > 75,000/mm3, total bilirubin < 2 mg/dl, serum creatinine < 2 mg/dl, Transaminases (AST, ALT) may be up to 2.0 x institutional upper limit of normal. In addition < 1 gr of protein in 24 hr urine collection and urine protein/creatinine ratio < 1.0.
* No life threatening parenchymal disease or rapidly progressing disease warranting cytotoxic chemotherapy.
* Hypertension must be controlled (<150/100 mmHg).
* Ejection Fraction > 50%.
* No history of thrombosis during the previous year.

Exclusion Criteria:

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than this sponsor-investigator Bevacizumab cancer study.
* Uncontrolled high blood pressure (150/100 mmHg)
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure see Appendix G)
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* History of a bleeding disorder
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein: creatinine ratio 1.0 at screening. Patients demonstrating > 1 gr of protein in 24 hr urine collection within 4 weeks prior to study entry will not participate in the trial.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Unwilling or unable to comply with the protocol for the duration of the study.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix.
* Patients with metastatic disease.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to estimate the pathological complete response rate of neoadjuvant therapy in operable newly diagnosed ER+ breast cancer patients using the combination of Avastin and Letrozole. | approximately 24 weeks

SECONDARY OUTCOMES:
A clinical response will be based upon the Response Evaluation Criteria in Solid Tumors (RECIST Criteria). | approximately 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andres Forero-Torres, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Vaklavas C, Roberts BS, Varley KE, Lin NU, Liu MC, Rugo HS, Puhalla S, Nanda R, Storniolo AM, Carey LA, Saleh MN, Li Y, Delossantos JF, Grizzle WE, LoBuglio AF, Myers RM, Forero-Torres A; Translational Breast Cancer Research Consortium (TBCRC). TBCRC 002: a phase II, randomized, open-label trial of preoperative letrozole with or without bevacizumab in postmenopausal women with newly diagnosed stage 2/3 hormone receptor-positive and HER2-negative breast cancer. Breast Cancer Res. 2020 Feb 18;22(1):22. doi: 10.1186/s13058-020-01258-x. PMID 32070401